CLINICAL TRIAL: NCT06544616
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blind, Parallel-Group Study, to Assess Efficacy, Safety and Immunogenicity of JNJ-64042056, a Phosphorylated Tau Targeted Active Immunotherapy, in Participants With Preclinical Alzheimer's Disease
Brief Title: A Study of JNJ-64042056 in Participants With Preclinical Alzheimer's Disease
Acronym: Reτain
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 64042056ALZ2001; 64042056ALZ2001 (Other: Janssen Research & Development, LLC); 2023-505096-68-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Preclinical Alzheimer's Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: JNJ-64042056 (Experimental): Participants will receive intramuscular (IM) injection of JNJ-64042056 from Week 0 until Week 180.
  Interventions: Drug: JNJ-64042056
- Arm B: Placebo (Placebo Comparator): Participants will receive IM injection of placebo from Week 0 until Week 180.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-64042056 — JNJ-64042056 will be administered intramuscularly.
  Arms: Arm A: JNJ-64042056
Drug: Placebo — Placebo will be administered intramuscularly.
  Arms: Arm B: Placebo

SUMMARY:
The purpose of this study is to assess the effect of JNJ-64042056 on cognitive decline, as measured by Preclinical Alzheimer's disease Cognitive Composite 5 (PACC-5) compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Elevated brain tau pathology defined as Braak 3 region of interest standardized uptake value ratio (ROI SUVR) greater than (>) 1.1 (or equivalent based on emerging data) on a screening tau PET scan, reviewed centrally by a qualified reader to enrich for probability of disease progression during the study
* Clinical Dementia Rating (CDR) global score of 0 at screening and baseline
* Mini Mental State Examination (MMSE) greater than or equal to (>=) 27 (with educational adjustment) at screening
* Able to read and write and with a minimum 5 years of formal education as reported by participant and study partner at screening
* A participant must be of non-childbearing potential

Exclusion Criteria:

* History consistent with or known autosomal dominant AD (mutation identified in the family and/or participant)
* Fulfills diagnostic criteria for Alzheimer's Dementia or non-Alzheimer's Dementia, including, but not limited to Frontotemporal Dementia (FTD), Diffuse Lewy Body Dementia (DLBD), Vascular Dementia (VAD), alcoholic dementia, Parkinson's dementia, Korsakov, Creutzfeldt-Jakob or other prion diseases, Posterior Cortical Atrophy
* Diagnosis of Mild Cognitive Impairment (MCI)
* Vitamin B12 or folate levels below the central laboratory lower limit of normal, unless the investigator determines that supplementation is not required after randomization
* History of or current neurological disease other than preclinical AD that may make interpretation of possible new neurological signs or symptoms difficult

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2031-07-17 (Estimated); Study Completion 2032-07-16 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Preclinical Alzheimer's Disease Cognitive Composite 5 (PACC-5) Total Scores up to Week 206 | Baseline up to Week 206
  Cognition will be measured using the PACC-5 scale, which includes 5 components: free/cued selective reminding test, delayed paragraph recall (logical memory test), digit-symbol substitution test, mini mental state examination, and the category fluency test (CFT). PACC-5 is a composite score which provides unique information about early cognitive decline not currently captured by the episodic memory, executive function, and global cognition components. The total score is a sum of z-score, with higher scores indicating better cognitive performance.

SECONDARY OUTCOMES:
Change From Baseline in Brain tau Burden as Measured by tau PET | Baseline and Weeks 102, 154 and 206
  Change from baseline in brain tau burden as measured by tau positron emission tomography (PET) at Weeks 102, 154 and 206 will be reported.
Change From Baseline in PACC-5 Individual Domain Scores | Baseline up to Week 206
  Cognition will be measured using the PACC-5 scale, which includes 5 components: free/cued selective reminding test, delayed paragraph recall (logical memory test), digit-symbol substitution test, mini mental state examination, and the category fluency test (CFT). PACC-5 is a composite score which provides unique information about early cognitive decline not currently captured by the episodic memory, executive function, and global cognition components. Each of the individual scales that are used to form PACC-5 composite score will be analyzed. Higher scores indicating better cognitive performance.
Time to Event of Clinical Progression as Measured by Clinical Dementia Rating-Global Score (CDR-GS) | Baseline up to Week 206
  Time to event of clinical progression as measured by clinical dementia rating-global score (CDR-GS) will be reported. The CDR assesses 3 domains of cognition (memory, orientation, judgment/problem solving) and 3 domains of function (community affairs, home/hobbies, personal care) using semi-structured interviews of both the study participant and the study partner carried out by a trained rater. Each domain is rated on a 5-point scale of functioning as follows: (0) no impairment; (0.5) questionable impairment; (1) mild impairment; (2) moderate impairment; and (3) severe impairment (Personal care is scored on a 4-point scale without a 0.5 rating available). CDR Global score ranging from 0 to 3, with 0 indicating no signs of clinically apparent cognitive impairment or dementia and 3 indicating severe dementia.
Change From Baseline in Clinical Dementia Rating-Sum of Boxes (CDR-SB) Scores | Baseline up to Week 206
  CDR assesses 3 domains of cognition (memory, orientation, judgment/problem solving) and 3 domains of function (community affairs, home/hobbies, personal care) using semi-structured interviews of both the study participant and the study partner carried out by a trained rater. Each domain is rated on a 5-point scale of functioning as follows: (0) no impairment; (0.5) questionable impairment; (1) mild impairment; (2) moderate impairment; and (3) severe impairment (Personal care is scored on a 4-point scale without a 0.5 rating available). Scores of the 6 domains (ranging from 0 to 3) summed to obtain the CDR. Sum of Boxes CDR-SB score with scores ranging from 0 to 18 where higher scores indicates greater impairment.
Change from Baseline in Tau PET Standardized Uptake Value Ratio (SUVR) Biomarkers | Baseline up to Week 206
  Change from baseline in Tau PET SUVR biomarkers will be reported.
Change From Baseline in p217+tau | Baseline up to Week 206
  Change from baseline in p217+tau will be reported.
Change From Baseline in PACC-5 Total Score | Baseline up to Week 180
  Change from baseline in PACC-5 total score will be reported.
Change From Baseline in Brain Tau Burden as Measured by Tau PET in Other ROI | Baseline up to Week 206
  Change from baseline in brain tau burden, as measured by tau PET (including but not limited to Braak I-VI ROIs, Connection Rank ROI, and New Tau Composite ROI Volume) will be reported.
Change From Baseline in Alzheimer's Disease Cooperative Study - Activities of Daily Living -Prevention Instrument (ADCS-ADL-PI) | Baseline up to Week 206
  The ADCS-ADL-PI is a functional measure composed of 18 items that include 15 activities of daily living rated on a 4-point scale and 3 high-level function items. Study participants and their study partners independently rate the participant's level of ability. Study partners are additionally asked to evaluate whether activities were completed less often, required more time to complete, and if any errors were made performing the task. High-level function items are rated as "yes" or "no". Total scores range from 0 to 45 with higher scores indicating less impairment.
Change From Baseline in Mild Behavioral Impairment Checklist (MBI-C) Score | Baseline up to Week 206
  MBI-C is a 2-page questionnaire consisting of 34 items, in 5 domains. The apathy domain consists of 6 questions including assessments of cognitive, behavioral and emotional apathy. The affect domain contains 6 items, including 4 for depressive features of low mood, anhedonia, hopelessness, and guilt, and 1 question each for worry and panic. The impulse dyscontrol domain is the largest, with 12 questions describing agitation, aggression, impulsivity, recklessness, and abnormal reward and reinforcement. The social appropriateness domain consists of 5 questions assessing sensitivity, empathy, and tact. Finally, the abnormal thought and perception domain consists of 5 questions assessing suspiciousness, grandiosity, and auditory and visual hallucinations.
Change From Baseline in the Quality of Life- Alzheimer's Disease (QoL-AD) | Baseline up to Week 206
  QoL-AD is a 13-item scale with four possible scores for each question (score 1: poor and score 4: excellent). It evaluates the caregiver's own perceived quality of life. Total score ranges from 13 to 52. Higher scores represent a better outcome.
Change From Baseline in European Quality of Life-5 Dimensions 5-Levels (EQ-5D-5L) Score | Baseline up to Week 206
  The EQ-5D-5L essentially consists of 2 elements: the European Quality of Life-5 Dimensions (EQ-5D) descriptive system and the European Quality visual analogue scale (EQ VAS). The EQ-5D descriptive system comprises the following 5 dimensions: mobility, selfcare, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and unable to/extreme problems. The digits for the 5 dimensions can be combined in a 5-digit number describing the respondent's health state which can be converted into a single summary index (EQ-5D index) by applying a formula that attaches values to each of the levels in each dimension. The EQ VAS records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labeled Best imaginable health state and Worst imaginable health state. The EQ VAS can be used as a quantitative measure of health outcome as judged by the individual respondents
Change From Baseline in Resource Utilization in Dementia-Lite (RUD-Lite) Score | Baseline up to Week 206
  RUD-Lite assesses the healthcare resource utilization of participants and their study partners and determines the level of formal and informal care attributable to Alzheimer's disease (AD). It assesses time spent in assisting participants with basics such as dressing, bathing and instrumental activities of daily living (ADLs) such as shopping and cooking. The RUD-Lite results can be used for calculating cost offsets and cost effectiveness modeling.
Levels of IgG Titers Against Enriched Paired Helical Filaments (ePHF), p-tau and tau in Serum | Up to Week 206
  Levels of IgG titers against ePHF, p-tau peptide and tau peptide in serum will be measured.
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Up to Week 208
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the pharmaceutical or biological agent under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Number of Participants With Reactogenicity | Up to Week 182
  Solicited AEs will be used to assess the reactogenicity of the active immunotherapy and are predefined local (at the injection site) and systemic events for which the participant is specifically questioned, and which are noted by participants in their participant diary.
Change from Baseline in Vital Signs | Baseline up to Week 180
  Change from baseline in vital signs including temperature and blood pressure (systolic and diastolic) (supine) will be summarized over time.
Change From Baseline in Clinical Laboratory Values | Baseline up to Week 206
  Change from baseline in clinical laboratory values (chemistry, hematology, urinalysis) will be reported.
Change from Baseline in Electrocardiogram (ECG) Values | Baseline up to Week 206
  Change from baseline in ECG values will be reported.
Change From Baseline in Columbia-Suicidality Severity Rating Scale (C-SSRS) | Baseline up to Week 206
  A frequency distribution of C-SSRS scores at each scheduled time point by treatment will be provided. Shifts from the baseline visit to the most severe/maximum score during the treatment period will be summarized by treatment. The maximum score assigned for each participant will also be summarized into 1 of 3 categories: no suicidal ideation or behavior (0), suicidal ideation (1 to 5), suicidal behavior (6 to 10).
Change From Baseline in Magnetic Resonance Imaging (MRI) Findings | Baseline up to Week 206
  Change from baseline in brain MRI safety findings will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V., Belgium Clinical trial, Study Director — Janssen Pharmaceutica N.V., Belgium
Locations (90):
- United States (34):
  - Xenoscience Inc., Phoenix, Arizona
  - Irvine Clinical Research, Irvine, California
  - Esperanza Clinical, Murrieta, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - JEM Research LLC, Atlantis, Florida
  - Excel Medical Clinical Trials, LLC, Boca Raton, Florida
  - K2 Medical Research Winter Garden, Clermont, Florida
  - Clinical NeuroScience Solutions Inc, Jacksonville, Florida
  - K2 Medical Research, Lady Lake, Florida
  - K2 Medical Research, Maitland, Florida
  - Merritt Island Medical Research, LLC, Merritt Island, Florida
  - Headlands Research Orlando, Orlando, Florida
  - Alzheimers Research and Treatment Center, Stuart, Florida
  - K2 Medical Research, Tampa, Florida
  - Charter Research, The Villages, Florida
  - Alzheimers Research and Treatment Center, Wellington, Florida
  - Palm Beach Neurology and Premier Research Institute, West Palm Beach, Florida
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Great Lakes Clinical Trials, Gurnee, Illinois
  - Quest Research Institute, Farmington Hills, Michigan
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - The Cognitive and Research Center of New Jersey LLC, Springfield, New Jersey
  - Neurological Associates of Albany, PC, Albany, New York
  - Velocity Clinical Research, East Syracuse, New York
  - The Medical Research Network, LLC, New York, New York
  - AMC Research, LLC, Matthews, North Carolina
  - Valley Medical Research, Centerville, Ohio
  - Keystone Clinical Studies LLC, Plymouth Meeting, Pennsylvania
  - Butler Hospital, Providence, Rhode Island
  - Clinical Trials of Texas Inc, San Antonio, Texas
  - Memory Clinic Inc, Bennington, Vermont
  - University of Virginia, Charlottesville, Virginia
- Australia (7):
  - Neuro Trials Victoria, Carlton
  - The Prince Charles Hospital, Chermside
  - St Vincent's Centre for Applied Medical Research, Darlinghurst
  - Austin Health Heidelberg Repatriation Hospital, Ivanhoe
  - Southern Neurology, Kogarah
  - KaRa Institute of Neurological Diseases, Macquarie Park
  - Australian Alzheimer's Research Foundation Incorporated, Nedlands
- Az Groeninge, Kortrijk, Belgium
- France (6):
  - Hopital Roger Salengro - CHU Lille, Lille
  - Hopital Nord Laennec CHU NANTES, Nantes
  - Hopital Lariboisiere-Fernand Widal, Paris
  - CHU Pitie Salpetriere, Paris
  - CHU Toulouse - Hôpital La Grave, Toulouse
  - CHRU Tours Hopital Bretonneau, Tours
- Germany (4):
  - Universitaetsklinikum der RWTH Aachen, Aachen
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum des Saarlandes, Homburg
  - Universitatsklinikum Munster, Münster
- Japan (13):
  - Enomoto Internal Medicine Clinic, Chofu-shi
  - Tokyo Asbo Clinic, Chūōku
  - Hatsuta Neurology Clinic, Hirakata-shi
  - Kobe City Medical Center General Hospital, Kobe
  - Kusunoki Clinic, Kobe
  - Musashimurayama Hospital, Musashimurayama
  - Saiseikai Narashino Hospital, Narashino-shi
  - ToCROM Clinic, Shinjuku Ku
  - Higashi-Shinjuku Clinic, Shinjuku-ku
  - Medical corporation Shinanokai Samoncho Clinic, Shinjyuku Ku
  - OCROM Clinic, Suita Shi
  - Nagomi Clinic, Toyonaka-shi
  - Jinsenkai MI Clinic, Toyonaka-shi
- Spain (11):
  - Barcelona Beta Brain Research Center, Barcelona
  - Fund. Ace-Inst. Cat. Neuroc. Aplicades, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Centro At. Esp. Oroitu, Getxo
  - Hosp. Univ. Santa Maria, Lleida
  - Hosp. Clinico San Carlos, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp. Quiron Madrid Pozuelo, Pozuelo de Alarcón
  - Idc Salud Hosp. Gral. de Catalunya, Sant Cugat del Vallès
  - Hosp. Mutua Terrassa, Terrassa
  - Hosp. Viamed Montecanal, Zaragoza
- Sweden (2):
  - Skanes universitetssjukhus, Malmo
  - Karolinska Universitetssjukhuset Huddinge, Stockholm
- United Kingdom (12):
  - Royal United Hospital, Bath
  - Re-Cognition Health, Birmingham
  - Re-Cognition Health, Bristol
  - Scottish Brain Sciences, Edinburgh
  - Re-Cognition Health, Guildford
  - Re-Cognition Health, London
  - Kings College Hospital, London
  - University of Oxford, Oxford
  - Re-Cognition Health, Plymouth
  - Moorgreen Hospital Memory Assessment And Research Centre, Southampton
  - Southampton General Hospital, Southampton
  - Re-Cognition Health, Winchester

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency